CLINICAL TRIAL: NCT01971554
Title: A Multiple Dose Clinical Trial to Study the Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of MK-8666 in Type 2 Diabetes Mellitus Patients
Brief Title: Safety, Tolerability, Pharmacodynamics, and Pharmacokinetics of MK-8666 in Participants With Type 2 Diabetes Mellitus (MK-8666-003)
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Merck Sharp & Dohme LLC (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 8666-003
Record Dates: First submitted 2013-10-14; First posted 2013-10-29 (Estimated); Results first posted 2016-12-08 (Estimated); Last update posted 2018-09-10 (Actual); Status verified 2018-08

CONDITIONS: Type 2 Diabetes Mellitus
MeSH Terms: conditions — Diabetes Mellitus, Type 2

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- MK-8666 50 mg (Experimental): MK-8666, 50 mg, oral, once a day (QD) for Days 1 to 14.
  Interventions: Drug: MK-8666; Drug: Placebo
- MK-8666 150 mg (Experimental): MK-8666, 150 mg, oral, QD, for Days 1 to 14
  Interventions: Drug: MK-8666; Drug: Placebo
- MK-8666 500 mg (Experimental): MK-8666, 500 mg, oral, QD for Days 1 to 14
  Interventions: Drug: MK-8666; Drug: Placebo
- Placebo (Placebo Comparator): Placebo, oral, QD for Days 1 to 14
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: MK-8666 — MK-8666, capsules, oral, QD, Days 1 to 14
  Arms: MK-8666 150 mg; MK-8666 50 mg; MK-8666 500 mg
Drug: Placebo — Placebo, capsules, oral, QD, Days 1 to 14

SUMMARY:
This is a study of the safety, tolerability, pharmacokinetics (PK), and pharmacodynamics (PD) of MK-8666 in participants with type 2 diabetes mellitus (T2DM). Participants enrolled in this trial would be either treatment-naive or have washed off of oral anti-hyperglycemic agents. MK-8666 is planned to be administered orally for up to 2 weeks. The primary hypothesis for this study is that after 14 days of once daily treatment with MK-8666, at a dose that is safe and well tolerated, the placebo-corrected fasting plasma glucose reduction from baseline is ≥34 mg/dL.

ELIGIBILITY:
Inclusion Criteria:

* If female, must be either postmenopausal or surgically sterile
* A Body Mass Index (BMI) ≥18 kg/m^2 to ≤40 kg/m^2, inclusive.
* A diagnosis of T2DM
* Drug naïve or is being treated with no more than 2 oral antihyperglycemic agents (thiazolidenediones are excluded)
* Judged to be in good health except for T2DM
* Willing to follow a standard weight maintaining diet throughout the study
* A nonsmoker or has not used nicotine or nicotine-containing products for at least 3 months

Exclusion Criteria:

* A history of clinically significant endocrine (except T2DM), gastrointestinal, cardiovascular, hematological, hepatic, immunological, renal, respiratory, or genitourinary abnormalities or diseases
* A history of myositis or complaints including diffuse myalgias, muscle tenderness, or weakness.
* A history of cancer (malignancy) excepting adequately treated non-melanomatous skin carcinoma or carcinoma in situ of the cervix
* Has clinically unstable diabetic retinopathy, neuropathy, and/or clinical evidence of gastroparesis (frequent nausea, bloating or vomiting, severe gastroesophageal reflux, early satiety)
* A history of type 1 diabetes mellitus and/or history of ketoacidosis
* Taking a medication for a co-morbid condition that is not permitted during the study
* A history of significant multiple and/or severe allergies
* Positive for hepatitis B surface antigen, hepatitis C antibodies or human immunodeficiency virus
* Had major surgery, donated or lost 1 unit of blood within 4 weeks prior to study participation
* Participated in another investigational trial within 4 weeks prior to study participation
* Consumes excessive amounts of alcoholic or caffeine-containing beverages
* A regular user of illicit drugs or a history of drug or alcohol abuse within the past year

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2013-10-14 (Actual); Primary Completion 2014-04-26 (Actual); Study Completion 2014-04-26 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Merck Sharp & Dohme LLC

IPD SHARING:
Plan to Share IPD: Yes
https://www.merck.com/clinical-trials/pdf/ProcedureAccessClinicalTrialData.pdf
URL: http://engagezone.msd.com/ds_documentation.php

REFERENCES:
- [Result] Krug AW, Vaddady P, Railkar RA, Musser BJ, Cote J, Ederveen A, Krefetz DG, DeNoia E, Free AL, Morrow L, Chakravarthy MV, Kauh E, Tatosian DA, Kothare PA. Leveraging a Clinical Phase Ib Proof-of-Concept Study for the GPR40 Agonist MK-8666 in Patients With Type 2 Diabetes for Model-Informed Phase II Dose Selection. Clin Transl Sci. 2017 Sep;10(5):404-411. doi: 10.1111/cts.12479. Epub 2017 Jul 20. PMID 28727908

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Sixty-three participants were recruited at 4 clinical sites in the United States.
Pre-assignment Details: Male and female participants with Type 2 diabetes mellitus between the ages of 18 and 65 years inclusive were enrolled in this trial.
Groups:
- MK-8666 50 mg: MK-8666 50 mg once daily for 14 consecutive days
- MK-8666 150 mg: MK-8666 150 mg once daily for 14 consecutive days
- MK-8666 500 mg: MK-8666 500 mg once daily for 14 consecutive days
- Placebo: Placebo once daily for 14 consecutive days
Period: Overall Study
Arm/Group | MK-8666 50 mg | MK-8666 150 mg | MK-8666 500 mg | Placebo
Started | 9 | 18 | 18 | 18
Completed | 8 | 18 | 18 | 18
Not Completed | 1 | 0 | 0 | 0
Not completed — Lost to Follow-up | 1 | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Total: Total of all reporting groups
Arm/Group | MK-8666 50 mg | MK-8666 150 mg | MK-8666 500 mg | Placebo | Total
Number analyzed (Participants) | 9 | 18 | 18 | 18 | 63
Age, Continuous [Mean (Full Range); unit: Years] | 53.9 (10.0) [30 to 65] | 55.6 (6.2) [46 to 65] | 55.2 (6.9) [37 to 64] | 54.7 (8.3) [36 to 64] | 55.0 [30 to 65]
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 4 | 6 | 7 | 8 | 25
  Male | 5 | 12 | 11 | 10 | 38

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Fasting Plasma Glucose (FPG) at Day 15
Description: Blood glucose was measured on a fasting basis (collected after an 8-hour fast). Blood was collected on Day -1 (pre-planned dose), predose on Days 1, 3, 7, and 14, and 24h postdose Day 14 (Day 15). The baseline measurement was computed as the average of the Day -1 and predose Day 1 measurements. FPG is expressed as mg/dL. This change from baseline reflects values for Day 15 FPG minus Day 0 FPG values.
Time Frame: Predose (Baseline) and 24 h postdose Day 14 (Day 15)
Population: The Per-Protocol population is the subset of participants who complied with the protocol sufficiently to ensure that these data are likely to exhibit the effects of treatment, according to the underlying scientific model.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | MK-8666 50 mg | MK-8666 150 mg | MK-8666 500 mg | Placebo
Number analyzed (Participants) | 9 | 18 | 18 | 18
mg/dL | 32.8 (9.7) | 37.9 (7.0) | 56.0 (7.0) | 2.0 (7.0)
Statistical Analysis 1: Comparison: MK-8666 50 mg vs Placebo; Test type: Superiority or Other; Difference in the least squares means = 30.8, 90% CI 2-sided [11.3 to 50.3] — A constrained longitudinal data analysis (cLDA) model was used to fit to the FPG data from the MK-8666 dose groups and placebo. Time was treated as a categorical variable so that no restriction was imposed on the trajectory of the means over time
Statistical Analysis 2: Comparison: MK-8666 150 mg vs Placebo; Test type: Superiority or Other; Difference in the least squares means = 36.0, 90% CI 2-sided [20.0 to 51.9] — A cLDA model was used to fit to the FPG data from the MK-8666 dose groups and placebo. Time was treated as a categorical variable so that no restriction was imposed on the trajectory of the means over time
Statistical Analysis 3: Comparison: MK-8666 500 mg vs Placebo; Test type: Superiority or Other; Difference in the least squares means = 54.1, 90% CI 2-sided [38.1 to 70.0] — [estimate comment as in outcome 1, analysis 2]

2. Primary Outcome: Number of Participants Who Experienced at Least Once Adverse Event
Description: An adverse event (AE) is defined as any unfavorable and unintended sign including an abnormal laboratory finding, symptom or disease associated with the use of a medical treatment or procedure, regardless of whether it is considered related to the medical treatment or procedure, that occurs during the course of the study.
Time Frame: Up to 28 days
Population: The Safety population consisted of all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | MK-8666 50 mg | MK-8666 150 mg | MK-8666 500 mg | Placebo
Number analyzed (Participants) | 9 | 18 | 18 | 18
Participants | 3 | 9 | 10 | 5

3. Primary Outcome: Number of Participants Who Discontinued Study Drug Due to an AE
Description: as for outcome 2
Time Frame: Up to 14 days
Population: The Safety population consisted of all participants who received at least one dose of study medication.
Measure: Number; unit: Participants
Arm/Group | MK-8666 50 mg | MK-8666 150 mg | MK-8666 500 mg | Placebo
Number analyzed (Participants) | 9 | 18 | 18 | 18
Participants | 0 | 0 | 0 | 0

4. Secondary Outcome: Area Under the Plasma Concentration-Time Curve From Time Zero to 24 Hours (AUC0-24h)
Description: AUC0-last is a measure of the total amount of drug in the plasma from the dose to 24 hours after the dose of study drug. Pharmacokinetic parameter analysis was not performed on the Placebo group. Method of dispersion for AUC0-24h was geometric mean coefficient of variation percentage.
Time Frame: Day 1: Predose, 0.5, 1, 1.5, 2, 2.5, 3, 4, 5, 6, 8, 12, 16, and 24 hours postdose; Day 14 : Predose, 0.5, 1, 2, 2.5, 3, 4, 6, 8, 12, 16, 24, 48, 72 hours postdose
Population: The Per-Protocol population is the subset of participants who complied with the protocol sufficiently to ensure that these data are likely to exhibit the effects of treatment, according to the underlying scientific model. Pharmacokinetic testing was not performed on the Placebo group.
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM·hr
Arm/Group | MK-8666 50 mg | MK-8666 150 mg | MK-8666 500 mg | Placebo
Number analyzed (Participants) | 9 | 18 | 18 | 0
μM·hr
  Day 1 | 6.11 (88) | 37.2 (44) | 143 (33) |
  Day 14 | 15.3 (88) | 66.9 (32) | 172 (37) |

5. Secondary Outcome: Maximum Plasma Drug Concentration After Dosing (Cmax)
Description: Cmax is a measure of the maximum amount of drug in the plasma after the dose of study drug. Pharmacokinetic parameter analysis was not performed on the Placebo group. Method of dispersion for Cmax was geometric mean coefficient of variation percentage.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Geometric Mean (Geometric Coefficient of Variation); unit: μM
Arm/Group | MK-8666 50 mg | MK-8666 150 mg | MK-8666 500 mg | Placebo
Number analyzed (Participants) | 9 | 18 | 18 | 0
μM
  Day 1 | 0.906 (102) | 4.49 (45) | 17.1 (40) |
  Day 14 | 1.50 (93) | 7.16 (37) | 19.9 (32) |

6. Secondary Outcome: Time to Reach Cmax (Tmax)
Description: Tmax is a measure of the time to reach the maximum concentration in the plasma after the dose of study drug. Pharmacokinetic parameter analysis was not performed on the Placebo group.
Time Frame: as for outcome 4
Population: as for outcome 4
Measure: Median (Full Range); unit: hr
Arm/Group | MK-8666 50 mg | MK-8666 150 mg | MK-8666 500 mg | Placebo
Number analyzed (Participants) | 9 | 18 | 18 | 0
hr
  Day 1 | 2.0 [1.5 to 12.0] | 2.25 [1.5 to 4.0] | 2.5 [1.5 to 8.0] |
  Day 14 | 2.0 [1.0 to 12.0] | 2.0 [1.0 to 6.0] | 2.0 [0.5 to 3.0] |

7. Secondary Outcome: Change From Baseline in 24-Hour Weighted Mean Glucose (24h-WMG) at Day 15
Description: The 24h-WMG was considered to provide an integrated assessment of the glycemic exposure over the 24-hour period, and was derived from 18 blood samples collected immediately prior to, and after each meal, and overnight and fasting one hour pre-dose. A "weighted" rather than a "simple" mean is used to avoid overrepresentation of post-meal glucose values. On each day (Day -1 and Day 14), the WMG was computed as a time-weighted average of the 18 individual measurements.
Time Frame: Baseline and Day 15
Population: The Per-Protocol population is the subset of participants who complied with the protocol sufficiently to ensure that these data are likely to exhibit the effects of treatment, according to the underlying scientific model. Data from 1 participant at Day 14 (Placebo group) was missing as the participant had to leave the study site.
Measure: Least Squares Mean (Standard Error); unit: mg/dL
Arm/Group | MK-8666 50 mg | MK-8666 150 mg | MK-8666 500 mg | Placebo
Number analyzed (Participants) | 9 | 18 | 18 | 17
mg/dL | 19.0 (7.9) | 27.3 (5.7) | 45.4 (5.7) | -3.3 (5.8)
Statistical Analysis 1: Comparison: MK-8666 50 mg vs Placebo; Test type: Superiority or Other; Difference in the least squares means = 22.3, 90% CI 2-sided [6.2 to 38.4] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 2: Comparison: MK-8666 150 mg vs Placebo; Test type: Superiority or Other; Difference in the least squares means = 30.6, 90% CI 2-sided [17.4 to 43.8] — [estimate comment as in outcome 1, analysis 2]
Statistical Analysis 3: Comparison: MK-8666 500 mg vs Placebo; Test type: Superiority or Other; Difference in the least squares means = 48.8, 90% CI 2-sided [35.6 to 62.0] — [estimate comment as in outcome 1, analysis 2]

ADVERSE EVENTS:
Time Frame: Up to 28 days
Arm/Group | MK-8666 50 mg | MK-8666 150 mg | MK-8666 500 mg | Placebo
Serious Adverse Events (participants affected / at risk) | 0/9 | 0/18 | 0/18 | 0/18
Other Adverse Events (participants affected / at risk) | 3/9 | 9/18 | 10/18 | 5/18
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | MK-8666 50 mg (N=9) | MK-8666 150 mg (N=18) | MK-8666 500 mg (N=18) | Placebo (N=18)
Bundle branch block right (Cardiac disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Eye irritation (Eye disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Eye redness (Eye disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Vision blurred (Eye disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Abdominal cramp (Gastrointestinal disorders) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Abdominal pain (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 0 (0)
Constipation (Gastrointestinal disorders) | 1 (1) | 3 (3) | 3 (4) | 1 (1)
Diarrhoea (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (2) | 1 (1)
Loose stools (Gastrointestinal disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Nausea (Gastrointestinal disorders) | 1 (1) | 0 (0) | 3 (4) | 1 (1)
Fatigue (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Upper respiratory tract infection (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Urinary tract infection (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Contusion of upper limb (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Post-traumatic pain (Injury, poisoning and procedural complications) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hyperglycaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 1 (2)
Back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Bone pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Flank pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 2 (2) | 0 (0)
Low back pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Neck pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Pain in foot (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pain in leg (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Shoulder pain (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 1 (3) | 0 (0)
Dizziness (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Drowsiness (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Drug-induced headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Headache (Nervous system disorders) | 2 (2) | 2 (2) | 3 (4) | 0 (0)
Occipital headache (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Urine discolouration (Renal and urinary disorders) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Rash maculo-papular (Skin and subcutaneous tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The sponsor must have the opportunity to review all proposed abstracts, manuscripts or presentations regarding this trial 45 days prior to submission for publication/presentation. Any information identified by the sponsor as confidential must be deleted prior to submission; this confidentiality does not include efficacy and safety results.